CLINICAL TRIAL: NCT05535595
Title: Precision Treatment Based on Genetic Information Associated With Response to Angiotensin Converting Enzyme Inhibitor
Brief Title: Precision Treatment With Angiotensin Converting Enzyme Inhibitor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-0916
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Genotype; Perindopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): This group will perform genetic study for predicting adverse reaction to ACEI. Based on the result of genetic study, participants will receive ACEI or ARB.
  Interventions: Drug: genotyping and selection of renin-angiotensin system blocker
- Control (Active Comparator): Participants will receive ACEI without genetic study.
  Interventions: Drug: Perindopril

INTERVENTIONS:
Drug: genotyping and selection of renin-angiotensin system blocker — One of perindopril or candesartan was chosen based on genotyping results on two NELL1 variants.
  * perindopril 4 mg/d after genotyping
  * candesartan 8 mg/d after genotyping
  Arms: Experimental
Drug: Perindopril — perindopril 4 mg/d without genotyping
  Arms: Control

SUMMARY:
Angiotensin converting enzyme inhibitors (ACEI) are the first-line treatment for high blood pressure and congestive heart failure, and have excellent effects in improving the prognosis of cardiovascular diseases. However, ACEI is frequently discontinued due to its adverse reaction. The adverse reaction to ACEI is not uncommon, especially in Asians. Discontinuation of ACEI is known to increase the risk of poor prognosis of cardiovascular diseases.

Biomarkers for predicting adverse reaction to ACEI have not yet been developed. Recently, genes related to adverse reaction to ACEI have been identified. This study is a randomized prospective study, in which the experimental group decides whether to administer the drug based on genetic information, and the control group decides whether to administer the drug without the information. In the experimental group, participants who are predicted to have a high risk of adverse reation to ACEI will receive angiotensin receptor blockers (ARB), and those who are predicted to have a low risk of adverse reaction will receive ACEI. Control group will receive ACEI. The frequency of adverse reaction will be investigated between control and experimental groups. In the genotyping and control groups, at least 45 and 31 will be enrolled, respectively, and after drug administration, a phone follow-up will be conducted at 3 weeks, followed by a visit at the 6th week, and the study will be terminated.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 20 years of age and less than 79 years of age
* Hypertension
* No history of ACEI use

Exclusion Criteria:

* Acute coronary syndrome, cerebrovascular accident, symptomatic peripheral artery disease, or coronary revascularization in the past three months
* Decompensated heart failure
* Systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg
* Hemoglobin A1c >9.0%
* Thyroid dysfunction
* Serum transaminase >2 times the upper limit of normal levels
* Serum creatinine >2.0 mg/dL
* Cancer
* Pregnant or breast-feeding women, and women of childbearing potential
* Patients who refused to participate

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Incidence of cough | 6 weeks after administration of drug
Incidence of moderate/severe cough | 6 weeks after administration of drug

SECONDARY OUTCOMES:
Incidence of any adverse events | 6 weeks after administration of drug

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hak Lee, Principal Investigator — Division of Cardiology, Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee SH, Lee CJ, Kang Y, Park JM, Lee JH. A randomized trial of genotype-guided perindopril use. J Hypertens. 2023 Nov 1;41(11):1768-1774. doi: 10.1097/HJH.0000000000003536. Epub 2023 Aug 17. PMID 37602458